CLINICAL TRIAL: NCT04218747
Title: Evaluation of Demonstrations to End Childhood Hunger - VA
Acronym: EDECHVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Food and Nutrition Service (U.S. Federal Agency)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-3198-C-14-0019 (Virginia)
Record Dates: First submitted 2019-12-12; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Food Insecurity Among Children
Keywords: Food Security; National School Lunch Program (NSLP); School Breakfast Program (SBP); Child and Adult Care Food Program (CACFP); Food Backpacks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA 365 Demonstration Benefits (Experimental): Children in treatment schools received: (1) three meals during the school day and food packages for weekends and school breaks; (2) $60 monthly Electronic Benefit Transfer (EBT) benefits during summer months if they were eligible for FRP meals; and (3) nutrition education for their parents.
  Interventions: Behavioral: VA 365 Demonstration Benefits
- Control Group (No Intervention): Schools in the control group operated under "business as usual."

INTERVENTIONS:
Behavioral: VA 365 Demonstration Benefits — Reducing hunger 365 days a year in households with school children by transforming schools into food hubs ( free breakfast, lunch, supper, and food backpacks for the weekend) and providing nutrition education to parents.
  Arms: VA 365 Demonstration Benefits

SUMMARY:
The 2010 Child Nutrition Reauthorization provided funding to test innovative strategies to end childhood hunger and food insecurity. Demonstration projects were funded in Chickasaw Nation, Kentucky, Navajo Nation, Nevada, and Virginia. This study focuses on Virginia. A selection of schools were randomly assigned to either a treatment or control group. Children in treatment schools received: (1) three meals during the school day and food packages for weekends and school breaks; (2) $60 monthly Electronic Benefit Transfer (EBT) benefits during summer months if they were eligible for FRP meals; and (3) nutrition education for their parents. The control group operated under "business as usual."

DETAILED DESCRIPTION:
Objective: To reduce hunger 365 days a year in households with schoolchildren by transforming schools into food hubs and providing nutrition education to parents.

Target Population: Elementary (n=30), middle (n=6), and high schools (n=2) in rural and urban VA. All schools had low academic performance and at least 50 percent of children eligible for free and reduced-price (FRP) meals.

Intervention: Schools were randomly assigned to either a treatment or control group. Children in treatment schools received: (1) three meals during the school day and food packages for weekends and school breaks; (2) $60 monthly Electronic Benefit Transfer (EBT) benefits during summer months if they were eligible for FRP meals; and (3) nutrition education for their parents. The control group operated under "business as usual." Note that the $60 monthly benefit was not included in the evaluation of the demonstration.

ELIGIBILITY:
Inclusion Criteria:

* A selection of elementary, middle, and high schools in rural and urban Virginia, USA.
* Schools must have had low academic performance and at least 50% or children eligible for free and reduced price through the National School Lunch Program or participating in the Community Eligibility Provision.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4750 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Food Insecurity among Children | Previous 30 days: once before intervention start and once during intervention implementation
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 2 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.

SECONDARY OUTCOMES:
Very Low Food Insecurity among Children | Previous 30 days: once before intervention start and once during intervention implementation
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 5 or more out of the 8 child-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Food Insecurity among Adults | Previous 30 days: once before intervention start and once during intervention implementation
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 10 adult-level items in the HFSSM. Higher scores generally indicates worsening food insecurity.
Household Food Insecurity | Previous 30 days: once before intervention start and once during intervention implementation
  Measured by the United States Department of Agriculture's Household Food Security Survey Module (HFSSM).
  Affirming 3 or more out of the 18 items in the HFSSM. Higher scores generally indicates worsening food insecurity.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Burke, PhD, Study Director — USDA Food and Nutrition Service

IPD SHARING:
Plan to Share IPD: Yes
Public-use data files are available by request by contacting Michael Burke (michael.burke@usda.gov) or the Office of Policy Support within the USDA Food and Nutrition Service.
URL: https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech

REFERENCES:
- See also: Final Report — https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech